CLINICAL TRIAL: NCT02238093
Title: Cardiorenal Syndrome in End-Stage Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 106-13-HYMC
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: End-stage Renal Disease; Cardiorenal Syndrome; Heart Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Cardio-Renal Syndrome; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dialysis Patients: End-stage renal disease patients undergoing dialysis at the Hillel Yaffe Medical Center.

SUMMARY:
Cardiorenal Syndrome (CRS) is prevalent among end-stage renal disease (ESRD) patients. Recently, its prevalence is rising. There are several different clinical presentations of this syndrome. It has a high rate of morbidity and mortality.

The purpose of this study is to find the connection between the heart pathology and its effect on ESRD patients. This will aid in choosing the appropriate medical therapy for these patients, and hopefully, aid in increasing their quality of life, and decrease their morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal patients

Exclusion Criteria:

* Cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients undergoing dialysis at the Hillel Yaffe Medical Center.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Heart Pathology Identification | One hour
  Visual identification of heart pathology in ESRD patients using echocardiography by measuring the ejection fraction of the left-ventricle during the systolic and diastolic phases. Valvular pathology is measured by the size of the valve.

CONTACTS AND LOCATIONS:
Overall Officials: Noa Berar-Yanay, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel